CLINICAL TRIAL: NCT06228885
Title: Investigating the Unique Motor Characteristics and Corresponding Cortical Activation During Handwriting -- in 5-12 Year-old Children With Autism Spectrum Disorder
Brief Title: Investigating Handwriting Characteristics and Underlying Factor in Children With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-111-277
Record Dates: First submitted 2023-12-27; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-12

CONDITIONS: Children With Autism Spectrum Disorder; Typical Developed Children
Keywords: Autism; Handwriting; Kinetic and kinematic; Cortical activation; Sensorimotor
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Autism Spectrum Disorder
  Interventions: Behavioral: handwriting experiment and motor ability test
- Typical developed children
  Interventions: Behavioral: handwriting experiment and motor ability test

INTERVENTIONS:
Behavioral: handwriting experiment and motor ability test — Participants will be instructed to participate in a handwriting experiment, which involves utilizing a Force Acquisition Pen (FAP) system and Near Infrared Spectroscopy (NIRS) to collect force data and cortical activation, respectively, during handwriting tasks. Children will be tasked with completing various assignments, such as tracing lines, writing numbers, and characters, among others. Additionally, assessments of motor ability and handwriting proficiency will be conducted using the Movement Assessment Battery for Children (MABC) and the Chinese Handwriting Evaluation Form (CHEF). The Pinch Holding Up Activity (PHUA) Test will also be administered to assess their sensorimotor ability.

SUMMARY:
The mechanism of the motor problem in children with autism spectrum disorder (ASD) in handwriting has been investigated in the following three aspects, including collecting dynamic handwriting performance, exploring the related underlying factors, and investigating corresponding brain activities. This study aimed to investigate the underlying factor of handwriting issue in children with ASD. There are four study aims. The first is to examine the differences of handwriting performance between children with ASD and TD using kinetic and kinematic measurements and handwriting difficulties questionnaires. The second is to investigate the group difference of the underlying motor factors, including fine motor ability and sensorimotor ability. The third is to explore the relationship between underlying motor factors and handwriting performance. The fourth is to explore the corresponding cortical activity during writing in children.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5-12 years old

Exclusion Criteria:

* who have a diagnosis of a seizure disorder, genetic condition, neurological condition, uncorrected significant hearing or visual impairment, and/or intellectual disability
* having non-verbal intelligent ability score lower than 70, determining by TONI-3
* unable to follow instructions during the process

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with ASD group:
  * Meeting the criteria for ASD according to DSM-5 from psychiatrist
  * ASD core symptoms: CARS higher than 30
  TD group:
  - The percentage score of MABC-2 is larger than 25% (not determined as "impaired motor coordination")
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Force-acquisition pen (FAP) system | baseline
  FAP system was used to collect the kinetic data during the process of writing. During the experiment, children will be asked to perform some tasks: tracing line, writing numbers, writing Bopomofo, and writing characters. The force of thumb, index, middle fingers and pen tip will be recorded. This is able to reflect the motor control aspect of handwriting through a variety of parameters. The following parameters will be calculated: average force, max force ration, numbers of force fluctuation per second, … and so on.
Pinch-Holding-Up Activity (PHUA) test | baseline
  The PHUA test is used to measure one's sensorimotor ability. Through calculating the parameters (max pinch force, max load force, force ratio … etc) to reflect one's ability to integrate sensory and produce a new output. A higher force ratio reflects a poorer sensorimotor ability.
Movement Assessment Battery for Children Second Edition (MABC-2) | baseline
  The MABC test is used to measure children's motor ability, including fine motor, balance and aiming and catching ability. The score will transform into z score and rank score, to reflect child's performance. A higher score indicates a better motor ability.
Chinese Handwriting Evaluation Form (CHEF) | baseline
  The CHEF is a questionnaire developed to assess and confirm the handwriting difficulties of preschooler (the third year of kindergarten) and school-aged children (grade one to two of elementary school). The school-aged version includes 25 items within five dimensions of handwriting problem: legibility, accuracy, speed, pencil grip, and directionality; while the preschooler version includes 22 items within four dimensions of handwriting problem: legibility, function (accuracy and speed), pencil grip, and attitude. The score is rated by teachers, parents, or familiar professionals with a 5-point Likert scale. A larger score indicates more difficulty in handwriting.

SECONDARY OUTCOMES:
Near Infrared Spectroscopy (NIRS) | baseline
  The NIRS system measures changes in oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR) as parameters to analyze cortical activation data. During handwriting, the cortical activation will be collected to observe which brain area activates more.

OTHER OUTCOMES:
Test of Nonverbal Intelligence, Third Edition (TONI-3) | baseline
  TONI is a test to evaluate one's nonverbal intelligence, without the influence of the confounding effects of linguistic or motor function. Children will conduct this test during screening phase.
Childhood Autism rating scale (CARS) | baseline
  CARS is a 15-items behavioral rating scale, for examining the autism symptoms in children. A higher score indicates more serious autistic symptoms. Parents will assist therapists in completing this scale during the screening phase.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided